CLINICAL TRIAL: NCT03874533
Title: Remote Monitoring Applied to Cochlear Implant Patient Follow-up (TELESURVIC)
Brief Title: Remote Monitoring Applied to Cochlear Implant Patient Follow-up
Acronym: TELESURVIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP180004
Record Dates: First submitted 2018-08-30; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Cochlear Diseases
Keywords: Cochlear Implantation; telemonitoring; training workshop
MeSH Terms: conditions — Cochlear Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- self-adjustment tests (Experimental): For patients with an implant Cochlear™, we will be trained during workshop, to use a tablet how to do some tests; They will do alone, by themselves the tests, just after the workshop and 8 to 30 days later.
  Self audiometric test : digit triplet test, consonants discrimination test, Self-fitting of cochlear implant
  Interventions: Device: Self-adjustment tests

INTERVENTIONS:
Device: Self-adjustment tests — For patients with an implant Cochlear™, we will be trained during workshop, to use a tablet how to do some tests ; They will do alone, by themselves the tests, just after the workshop and 8 to 30 days later.
  Self audiometric test : digit triplet test, consonants discrimination test, Self-fitting of cochlear implant

SUMMARY:
The cochlear implant (CI) is a device to compensate severe or profound deafness. The CI has a lifetime implanted part and an external processor. Regular monitoring is necessary because the device can generate complications and when the device is dysfunctional, the patient becomes deaf again. Our center, the CRIC, is a center for monitoring and fitting CI. Follow-up requires face-to-face procedures and some patients have difficulty accessing the center.

Our cohort of patients is growing steadily and now exceeds 750 patients. Provision should be made for sustained steady growth and enabling means. Telemedicine may be a response for the follow-up of some patients.

Currently, cochlear implanted patients benefit once a year from: an ENT (Ear Nose and Throat) medical consultation, a speech-language assessment, physical verification of the external processor, an audiometric test, a fitting of the external processor. This makes it possible to check the absence of medical complication, the use and the correct functioning of the external and internal parts.

Provision should be made for sustained steady growth and enabling means. With the development of new hearing tests, technical possibilities of some speech processors and software for their fitting, telemedicine may be a response for the follow-up of some patients.

TELESURVIC will study the feasibility for patients implanted with an implant Cochlear™ to carry out a complete test of their equipment by themselves.

For this project we will use a tablet device, without simultaneous contact with CRIC professionals. On this tablet are installed calibrated hearing tests, tutorials of good maintenance of the processor and a software of adjustment allowing the realization of the operations desired for an inspection of the implant.

Patients selected to participate, (on a voluntary basis), in this protocol will follow the following steps:

1. They will first be trained in the use of the tablet at the CRIC by professionals. Patients will only be included if they are autonomous in handling the tablet and specific software;
2. They will carry out the various tests at the hospital on the tablet: audiometry test in quiet and in noise then checking of the data logging, self-fitting thanks to the Cochlear software (NFS);
3. Between one week and one month later, they will come back to the center and will do the same tests alone in a quiet room of the center.
4. Outside the patient's presence, the data will be analyzed and compared with the data collected in step 2, in order to validate or not, the feasibility of these self-administrated tests without any help by the team.

DETAILED DESCRIPTION:
The selection of the patients is made on study of the files of the cochlear implanted patients with leading implant COCHLEARTM, compatible external processor with the research and being able to potentially realize only the studied acts.

The unit proposes then during a consultation or by explanatory e-mail, to the patient to participate in a training workshop. The information note will be presented to the patient during the consultation, or sent by e-mail.

After checking the selection criteria and signing the consent by the patient, the patient joins a training workshop.

During the workshop, bringing together 3 to 5 patients supervised by an ENT doctor of the +/- adjuster team, a speech therapist and +/- a COCHLEARTM engineer, patients will be trained in the handling of the tablet and software. Then, in a second step, each patient will have to carry out the hearing and self-adjustment tests by themselves in a quiet room in the unit. He will be able to reach a unit professional who can help him.

The patient will benefit from auditory evaluation by a consonants discrimination test and a 3-digit noise test and then an evaluation of the implant and processor parameters using COCHLEARTM NFS tuning software.

It is at the end of this workshop that the unit professionals will judge whether the patient is pursuing the research or not. If the patient continues the research, he will have an appointment to return to the service 8 to 30 days later.

Patients pursuing the research will be invited to complete the end-of-workshop questionnaire.

The patient will return to the follow-up center and will repeat exactly the same acts, alone in a room, 8 to 30 days after the first tests. He will also have the opportunity to be assisted by someone of his choice.

At the end of this visit, the patient will be invited to complete the end-of-research questionnaire.

This follow-up visit will mark the end of the patient's participation in this research, unless there is a need to adjust the device.

Once the tests are completed, health professionals will analyze the data retrieved from the tablet and if needed, will see the patient in adjustment within 8 days maximum if there is a difference between the tests performed at the unit during the inclusion visit and those performed by the patient alone in a distant evaluation.

Self-test data from the patient at the follow-up visit should be identical to the training workshop. If this is not the case, it is therefore essential to know if the difference is due to a poor control of the tests or rather to an anomaly appeared secondarily.

Patients will be reviewed as part of the care in case of need for new settings.

The professionals involved in the research (training workshop and self-test verification) will be invited to complete an evaluation questionnaire

Our approach aims to make the patient aware of how the cochlear implant works, to empower him and to make him responsible for his equipment.

By providing him with training not only in passing evaluation self-tests but also in certain parameters of the setting, we want him to understand the interest of an annual follow-up.

And we want to show that a well-trained patient can participate actively in the follow-up of his cochlear implant thanks to adapted tools and telemedicine.

Total number of subjects selected to participate in the workshop: 40. Inclusion period: 6 months, for 30 selected patients at the end of the workshop.

Duration of participation of each patient: 38 days maximum Total search time: 7 months and 8 days

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old
* Cochlear implantation older than 6 months (with a COCHLEAR implant and processor allowing wireless connection), followed by CRIC or IFIC,
* Fluent in the French language,
* Possibility of carrying out the acts alone in person in the service within a short time (less than 30 days).
* Patients affiliated to a social security scheme or entitled to it
* Patient who has signed informed consent form

Exclusion Criteria:

* Difficulty mastering the tests alone or handling the tablet that will be entrusted to him
* Persons deprived of their liberty by judicial or administrative decision
* Persons hospitalized without consent and without legal protection, and persons admitted to a health or social institution for purposes other than research.
* Adults who are subject to a legal protection measure (guardianship, trusteeship or judicial protection), adults who are unable to express their consent and are not subject to a protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The degree of auditory rehabilitation achieved with the cochlear implant. | Between day +8 to +30 after the training session
  Comparison of the data collected (The hearing tests 3 digits test and VCV) during the usual evaluations in the department, then in auditory self-test and of the parameters of reaction just after an apprenticeship and at a distance, between 8 to 30 days, of this learning
The degree of auditory rehabilitation achieved with the cochlear implant. | Between day +8 to +30 after the training session
  Comparison of the data collected (the electrophysiological measures) during the usual evaluations in the department, then in auditory self-test and of the parameters of reaction just after an apprenticeship and at a distance, between 8 to 30 days, of this learning

SECONDARY OUTCOMES:
Estimate the degree of patients satisfaction, on the use of new tools that will be used for remote monitoring | Between day +8 to +30 after the training session
  For the patients: The results of Qualitative Self questionnaire, EVA scale, and free comments, according to the scoring manual, will be aggregated to estimate the degree of satisfaction.
Estimate the degree of satisfaction professionals, on the use of new tools that will be used for remote monitoring | Between day +8 to +30 after the training session
  For the professionals: The results of Qualitative Self questionnaire, EVA scale, and free comments, according to the scoring manual, will be aggregated to estimate the degree of satisfaction.
Estimate the necessary adaptations of the medical team and patients | Between day +8 to +30 after the training session
  When the patients come back (between Day +8 to Day+30), they do the same tests alone, by themselves. The staff checks if the results are the same as those of the tests at day 0, (without any medical or technical intercurrent event).
  We note the time spent for each test by the patient. Each professional involved in the process of teaching, coaching and assessing the patient through the study will fill a chart detailing his/her actions and keep a record of his/her dedicated time.
  By this approach, we hope building a team adapted to the remote monitoring applied to cochlear implant patient follow-up.
Estimate time savings for professionals | Between day +8 to +30 after the training session
  Comparison of the time spent for acts realized in a traditional way and the way according to the protocol, for professionals.
Estimate time savings for patients | Between day +8 to +30 after the training session
  Comparison of the time spent for acts realized in a traditional way and the way according to the protocol, for patients.

CONTACTS AND LOCATIONS:
Overall Officials: Christine PONCET WALLET, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No